CLINICAL TRIAL: NCT04434911
Title: Precision Medicine Study on Cardiovascular Disease (PRECISE)
Acronym: PRECISE
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei.Song@NCCD, Principal Investigator, China National Center for Cardiovascular Diseases
Other Study IDs: PRECISE
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
Keywords: monogenic cardiovascular disease; clinical outcomes; genomics; genetic diagnosis; risk stratification
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Specimens retained include blood, saliva, urine, feces, and myocardium when the patients receive cardio myectomy surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular diseases are the leading cause of death in China and have become a financial burden on society under the traditional medical model. A new and sustainable medical model is needed to solve this dilemma, for which precision medicine models have great potential. Monogenic cardiovascular disease is the first field to be broken through in precision medicine at this stage, and it is also the field where precision medicine is most likely to be successfully transformed into clinical application, including genetic diagnosis, molecular typing, risk stratification, genetic interruption and individualized treatment.

DETAILED DESCRIPTION:
In this study, patients with monogenic cardiovascular disease are recruited prospectively after informed consent was given. The investigator will collect the baseline clinical characteristics of the patients at enrollment, including comprehensive physical examination, laboratory testing of blood and urine, electrocardiography, 24-hour Holter, echocardiography, MRI and other examinations if necessary. The specimens retained include blood, saliva, urine and feces for all patients, and myocardium for patients receive cardio myectomy surgery . Genetic testing will be performed to identify novel disease genes, genetic risk factors and potential therapy targets.

ELIGIBILITY:
Inclusion Criteria:

* Patients with monogenic cardiovascular diagnosed according current practice guideline.

Exclusion Criteria:

* Patients who refuse to sign the informed consent or decline follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with monogenic cardiovascular disease from multiple centers in China between October 10, 2020 and October 10, 2025
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
number of participants with cardiovascular deaths | an average of 5 years
  including sudden cardiac death and deaths due to heart failure and stroke.
number of participants with all-cause death | an average of 5 years.
  deaths due to all cause.

SECONDARY OUTCOMES:
number of participants with heart failure | an average of 5 years
  progress to level III or IV in New York Heart Association class.
number of participants with stroke | an average of 5 years
  including cerebral infraction and hemorrhage
number of participants with malignant arrhythmia | an average of 5 years
  including ventricular fibrillation and ventricular tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Lei Song, MD. ph.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided